CLINICAL TRIAL: NCT00049348
Title: A Randomized Phase II Study Of Gemcitabine Plus Radiotherapy Vs. Gemcitabine, 5-Fluorouracil And Cisplatin Followed By Radiotherapy And 5-Fluoraracil For Patients With Locally Advanced, Potentially Resectable Pancreatic Adenocarcinoma
Brief Title: Chemotherapy and Radiation Therapy in Treating Patients With Locally Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Group Chair, Eastern Cooperative Oncology Group
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000258056; E1200
Record Dates: First submitted 2002-11-12; First posted 2003-01-27 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage II pancreatic cancer; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Epoetin Alfa; Filgrastim; Cisplatin; Fluorouracil; Gemcitabine; Chemotherapy, Adjuvant; Neoadjuvant Therapy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: epoetin alfa
Biological: filgrastim
Drug: cisplatin
Drug: fluorouracil
Drug: gemcitabine hydrochloride
Procedure: adjuvant therapy
Procedure: conventional surgery
Procedure: neoadjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy before surgery may shrink the tumor so that it can be removed during surgery.

PURPOSE: Randomized phase II trial to compare the effectiveness of two different regimens combining chemotherapy with radiation therapy in treating patients who are undergoing surgery for locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the percentage of margin-free resections in patients with locally advanced, potentially resectable adenocarcinoma of the pancreas treated with gemcitabine and radiotherapy vs gemcitabine, fluorouracil, and cisplatin followed by radiotherapy and fluorouracil.
* Compare the efficacy of these regimens, as measured by CT scan response, in these patients.
* Compare the posttreatment fibrosis in resected specimens of patients treated with these regimens.
* Compare the toxicity of these regimens in these patients.
* Compare the duration of objective response in patients treated with these regimens.
* Compare the disease-free and overall survival of patients treated with these regimens.
* Compare the effect of these regimens and disease recurrence on CA 19-9 values in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to superior mesenteric vein (SMV)/portal vein (PV) occlusion (yes vs no), SMV/PV/superior mesenteric artery/hepatic artery abutment or narrowing (yes vs no), prior exploration (yes vs no), and whether deemed to require preoperative therapy due to other factors (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo radiotherapy once daily 5 days a week for 6 weeks. Patients receive gemcitabine IV over 50 minutes once weekly for 6 weeks during radiotherapy. Patients undergo surgical resection 4-6 weeks after completion of chemoradiotherapy.

Maintenance therapy (4-8 weeks after completion of surgery): Patients receive gemcitabine IV over 100 minutes once weekly for 2 weeks. Treatment repeats every 3 weeks for 5 courses in the absence of disease progression or unacceptable toxicity.

* Arm II: Patients receive gemcitabine IV over 30 minutes on days 1, 5, 29, and 33; cisplatin IV over 60 minutes on days 1-5 and 29-33; and fluorouracil IV continuously on days 1-4 and 29-32. Patients also receive filgrastim (G-CSF) subcutaneously (SC) daily on days 6-15 and 34-43 and epoetin alfa SC weekly on weeks 1-9. After completion of chemotherapy, patients undergo radiotherapy once daily 5 days a week for 6 weeks. Patients receive fluorouracil IV continuously daily during radiotherapy. Patients undergo surgical resection 4-6 weeks after completion of chemoradiotherapy.

Maintenance therapy (4-8 weeks after completion of surgery): Patients receive gemcitabine IV over 100 minutes once weekly for 2 weeks. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 80-160 patients (40-80 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the pancreas

  * No adenosquamous cancers or adenocarcinoma associated with cystic mucinous neoplasms
  * Locally advanced disease that is potentially resectable, previously explored and considered unresectable, or deemed to require preoperative treatment for other reasons
  * Primary cancer in the head, body, or tail of pancreas
* Measurable disease
* No 360 degree encirclement of the superior mesenteric artery, hepatic artery, or celiac axis
* No metastases by CT scan and laparoscopy (if prior surgery, only CT scan required)

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count greater than 2,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* Bilirubin less than 2 mg/dL (unless secondary to bile duct blockage by tumor)
* Biliary obstruction by tumor requires biliary stent at least 9 French or biliary bypass before therapy

Renal

* Creatinine less than 1.7 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Other

* No other malignancy within the past 3 years except nonmelanoma skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for this disease

Endocrine therapy

* Not specified

Radiotherapy

* No prior radiotherapy to pancreas

Surgery

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-10-13 (Actual); Primary Completion 2005-10 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Percentage of margin-free resections produced by each program

SECONDARY OUTCOMES:
Efficacy as measured by CT scan response
Post-treatment fibrosis in the resected specimens
Toxicity
Duration of objective response
Disease-free survival
Overall survival
Effect of therapy and recurrence on CA19-9 values

CONTACTS AND LOCATIONS:
Overall Officials: John Parker Hoffman, MD, Study Chair — Fox Chase Cancer Center
Locations (137):
- United States (137):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Lynn Regional Cancer Center of Boca Raton Community Hospital, Boca Raton, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Veterans Affairs Medical Center - Lakeside Chicago, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - St. Anthony's Memorial Hospital, Effingham, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Evanston Northwestern Health Care - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - InterCommunity Cancer Center of Western Illinois, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Joliet Oncology Hematology Associates, Limited - West, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - Deerpath Medical Associates, Lake Forest, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Northwest Medical Specialist P.C., Niles, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois - Ottawa, Ottawa, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Hematology Oncology Associates - Skokie, Skokie, Illinois
  - Hematology/Oncology of the North Shore, Skokie, Illinois
  - Midwest Cancer Research Group, Incorporated, Skokie, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Valley Cancer Center, Spring Valley, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Saint Joseph Regional Medical Center - Plymouth Campus, Plymouth, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - McFarland Clinic, P.C., Ames, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology-Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, P.A. - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Cancer Center of Kansas - Ottawa, Ottawa, Kansas
  - Cancer Center of Kansas, P.A. - Parsons, Parsons, Kansas
  - Pratt Cancer Center of Kansas, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates in Womens Health, Wichita, Kansas
  - Cancer Center of Kansas, P.A., Wichita, Kansas
  - Cancer Center of Kansas, P.A. - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Baton Rouge General Regional Cancer Center, Baton Rouge, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Cancer Center at Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Franklin Medical Center, Greenfield, Massachusetts
  - Holyoke Medical Center, Incorporated, Holyoke, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Noble Hospital, Westfield, Massachusetts
  - MeritCare Clinic - Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Mercy and Unity Hospitals, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Clinic, Saint Louis Park, Minnesota
  - Cancer Care Center at Regions Hospital, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Woodwinds Hospital, Woodbury, Minnesota
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Health System, Bismarck, North Dakota
  - Mid Dakota Clinic, P.C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Medical Group, Fargo, North Dakota
  - St. Elizabeth Boardman Cancer Center, Boardman, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - St. Joseph Health Care Center, Warren, Ohio
  - St. Elizabeth Cancer Center at St. Elizabeth Health Center - Youngstown, Youngstown, Ohio
  - St. Luke's Hospital Cancer Center, Bethlehem, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Avera McKennan Hospital and University Health Center, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Erlanger Cancer Center, Chattanooga, Tennessee
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin

REFERENCES:
- [Result] Landry JC, Catalano P, Hoffman J, et al.: ECOG 1200: a randomized phase II trial of gemcitabine plus radiotherapy vs gemcitabine, 5-fluorouracil and cisplatin followed by radiotherapy and 5-fluorouracil in patients with locally advanced, potentially resectable pancreatic adenocarcinoma. [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-2111, S272, 2006.